CLINICAL TRIAL: NCT01346072
Title: Pilot Study of the Relationship of Ambient Copeptin to the Aquaretic Effects of Tolvaptan in Patients With Heart Failure
Brief Title: Pilot Study of Using Copeptin to Predict Response to Tolvaptan
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Otsuka America Pharmaceutical (Industry)
Responsible Party: Principal Investigator, Kirkwood Adams, Associate Professor of Medicine and Radiology, University of North Carolina, Chapel Hill
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TOLCOPEP11
Record Dates: First submitted 2011-04-29; First posted 2011-05-02 (Estimated); Results first posted 2017-05-17 (Actual); Last update posted 2017-05-17 (Actual); Status verified 2017-04

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Heart Failure
Keywords: tolvaptan; copeptin; heart failure; vasopressin antagonist
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Heart Failure; Diabetes Insipidus | interventions — Tolvaptan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tolvaptan (Other): Single arm study
  Interventions: Drug: tolvaptan

INTERVENTIONS:
Drug: tolvaptan — oral, 30 mg, single dose, one time administration
  Other Names: Samsca

SUMMARY:
This pilot study will investigate the association between levels of the peptide copeptin and response to tolvaptan, a drug that blocks the action of the water retaining hormone vasopressin. The study will enroll stable outpatients with CHF with reduced LVEF (≤45) selected by targeting upper and lower quartile copeptin levels at screening (10 each). The treatment phase of the study will be a prospective, single-arm, open label protocol. All patients will receive active therapy consisting of a single oral dose of 30 mg of tolvaptan with body weight, fluid intake, and urine output monitored in a research unit for 24 hours.

For analysis of study endpoints, patients in the single intervention arm will be stratified by a prospectively determined cut-point of copeptin level into two groups (≥10 versus <10 pmol/L). The copeptin level used for the two group stratification will be the blinded copeptin value obtained at baseline from the hospital phase prior to administration of tolvaptan.

DETAILED DESCRIPTION:
The study screening strategy will be designed to enroll an enriched patient population by identifying patients at the high or low end of the spectrum of copeptin levels for outpatients with stable heart failure. This will be accomplished by blinded review of copeptin levels obtained during screening.

The primary endpoints for analysis will be 24 hour urine output and the change in body weight over 24 hours during the inpatient stay.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients with a history of chronic symptomatic heart failure, defined as dyspnea on exertion or edema, due to cardiac dysfunction, of at least one month's duration
2. Left ventricular ejection fraction ≤ 45% as documented by quantitative assessment by an accepted imaging technique within one year of screening
3. Meet baseline copeptin criteria for entry
4. Currently taking a diuretic (with diuretic defined as any loop or thiazide diuretic or aldosterone antagonist at any dose)

Exclusion Criteria:

1. Current New York Heart Association Functional Class IV heart failure
2. Patients who are felt to be volume depleted based on clinical examination or need to reduce diuretic administration
3. Presence of clinical contraindications to tolvaptan
4. Episode of acute myocardial infarction or acute coronary syndrome within the past 3 months
5. Cardiovascular surgical procedure within the past 4 weeks
6. CHF due to uncorrected thyroid disease, active myocarditis, or known amyloid cardiomyopathy.
7. History of primary significant liver disease or acute hepatic failure, as defined by the investigator.
8. Chronic uncontrolled diabetes mellitus as determined by the investigator.
9. Supine systolic arterial blood pressure < 90 mmHg at screening
10. Serum creatinine > 3.5 mg/dL at screening
11. Serum potassium > 5.5 mEq/L or < 3.5 mEq/L at screening
12. Subjects currently treated with hemofiltration or dialysis

j. Subjects judged by the investigator to be unable to maintain accurate intake and output during their hospitalization related to medical or other problems

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2011-04; Primary Completion 2014-02 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kirkwood F Adams, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 100 patients were screened in two periods approximately six months each in duration at a dedicated Heart Failure Clinic at the University of North Carolina Chapel Hill. 43 patients met inclusion/exclusion criteria and had a blood sample sent for copeptin testing. Twenty-one patients were enrolled in the hospital phase of the study.
Pre-assignment Details: Blinded copeptin results were reviewed in 43 patients for participation in the hospital phase. 11 patients were selected by targeting the upper quartile of baseline copetin and 10 patients by targeting the lower quartile of screening copeptin levels. A total of 21 patients were enrolled in hospital phase.
Groups:
- Tolvaptan High Copeptin: Tolvaptan: oral, 30 mg, single dose, one time administration
  High Copeptin ≥ 10 pmol/L at baseline
- Tolvaptan Low Copeptin: Tolvaptan: oral, 30 mg, single dose, one time administration
  Low Copeptin < 10 pmol/L at baseline
Period: Overall Study
Arm/Group | Tolvaptan High Copeptin | Tolvaptan Low Copeptin
Started | 11 | 10
Completed | 11 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All patients in Low Copeptin group were included in analysis. One patient in High Copeptin group had reduced renal function at baseline versus screening and transient hypovolemia during hospitalization indicative of volume depletion. This patient was excluded prior to review of blinded copeptin results and study data analysis for a final N of 20.
Groups:
- Total: Total of all reporting groups
Arm/Group | Tolvaptan High Copeptin | Tolvaptan Low Copeptin | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 7 | 14
  >=65 years | 3 | 3 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 60 (11) | 59 (13) | 60 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 11
  Male | 5 | 4 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 4 | 11
  White | 3 | 5 | 8
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20
LVEF [Mean (Standard Deviation); unit: %] | 23 (6.0) | 31 (11) | 27 (9.6)
Baseline Copeptin [Mean (Standard Deviation); unit: pmol/L] | 20.5 (8.7) | 5.7 (1.9) | 13.1 (9.7)
Serum Creatinine [Mean (Standard Deviation); unit: mg/dL] | 1.18 (0.23) | 1.03 (0.35) | 1.10 (0.30)
Serum Sodium [Mean (Standard Deviation); unit: mEq/L] | 141.1 (2.28) | 140.8 (3.46) | 141.0 (2.86)
Total Daily Dose of Loop Diuretic [Mean (Standard Deviation); unit: mg] | 124 (104) | 47 (46) | 84 (86)

OUTCOME MEASURES:

1. Primary Outcome: Urine Output
Description: Total urine output for 24 hours following tolvaptan administration
Time Frame: 24 hours
Population: All patients in the Low Copeptin group were included in the analysis. One patient in the High Copeptin group had reduced renal function at baseline versus screening and transient hypovolemia during hospitalization indicative of volume depletion. This patient was excluded prior to review of blinded copeptin results and study data analysis.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Tolvaptan High Copeptin | Tolvaptan Low Copeptin
Number analyzed (Participants) | 10 | 10
mL | 6498 (2328) | 5784 (1835)
Statistical Analysis 1: Comparison: Tolvaptan High Copeptin vs Tolvaptan Low Copeptin; Test type: Superiority; p = 0.853, Wilcoxon Two-Sample Test; Wilcoxon Two Sample Test was used with Exact Test two sided p value reported

2. Primary Outcome: Body Weight
Description: Change in body weight from baseline to 24 hours after tolvaptan administration
Time Frame: Change over 24 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Kg
Arm/Group | Tolvaptan High Copeptin | Tolvaptan Low Copeptin
Number analyzed (Participants) | 10 | 10
Kg | -1.3 (1.0) | -0.4 (1.0)
Statistical Analysis 1: Comparison: Tolvaptan High Copeptin vs Tolvaptan Low Copeptin; Test type: Superiority; p = 0.035, Wilcoxon Two-Sample Test; Wilcoxon Two Sample Test was used with Exact Test two sided p value reported

ADVERSE EVENTS:
Time Frame: 24 hours
Arm/Group | Tolvaptan High Copeptin | Tolvaptan Low Copeptin
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/10
Other Adverse Events (participants affected / at risk) | 0/11 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less